CLINICAL TRIAL: NCT00147394
Title: Risperidone Pharmacokinetics in Children With Pervasive Developmental Disorder
Brief Title: Risperidone Pharmacokinetics in Children With Pervasive Developmental Disorder (PDD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPRU 10544
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Child Development Disorders, Pervasive
Keywords: Risperidone; Autism; PDD; Pervasive Developmental Disorder
MeSH Terms: conditions — Child Development Disorders, Pervasive; Autistic Disorder | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this research is to study the pharmacokinetics of risperidone in a group of pediatric patients with Pervasive Developmental Disorder (PDD). The study will determine how much risperidone and its breakdown product, 9-hydroxy-risperidone, is in the blood following the patient's usual daily dose. The study is designed to look at how fast children absorb, breakdown, and eliminate risperidone.

DETAILED DESCRIPTION:
Pervasive Developmental Disorders is a category of disorders that includes autism and related conditions. While these disorders are rare, they represent a significant public health problem because they are extremely debilitating and lack efficacious therapies. Neuroleptic use in PDD is high and the population appears to be at increased risk of serious sequelae including tardive dyskinesia. Newer atypical neuroleptics including risperidone are now used in 87% of cases but dosing, safety and efficacy is undetermined in the vulnerable population.

This study consists of a total of 3 visits, the initial screening visit where consent, medical history, demographics and vitals will be recorded. Two additional visits with blood sampling will occur. The second visit will be no greater than 30 days from the screening visit and the 3rd visit will be one month from Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between ages of 5 and less than 17 years.
* Patients meeting DSM-IV criteria for PDD-NOS about to initiate clinical treatment or currently clinically treated with risperidone.
* Patients with autistic disorder or PDD-NOS currently on risperidone as a participant in one of the multi-site RUPP protocols.

Exclusion Criteria:

* Children taking psychotropic or other medication that will interact with target CYP 450 isoenzyme activity will not be eligible for the pharmacokinetic study (i.e. CYP2D6 or CYP3A4; to be decided by the PI)
* Patients with known renal or hepatic dysfunction (e.g. serum creatinine > 1.5 normal upper limit, transaminases or bilirubin > 2 times normal upper limit)
* Failure of the parent/legal guardian to give informed consent.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2001-12; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Quantify the variability of clearance and volume of distribution among AE rating, weight gain and ABC responder status.

SECONDARY OUTCOMES:
Exploratory analysis will be performed to examine the relationship of other factors to risperidone and metabolite concentrations for PK/PD assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Vinks, Pharm.D., Ph.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (5):
- United States (5):
  - Children's Hospital of Michigan/Wayne State University, Detroit, Michigan
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio